CLINICAL TRIAL: NCT07042529
Title: Optimized Expansion of the Implanted Transcatheter Aortic Valve to Reduce Hypoattenuating Leaflet Thickening in Non-atrial Fibrillation Patients Undergoing Transcatheter Aortic Valve Implantation: an International, Multicentre, Randomized Controlled Trial
Brief Title: Optimized Expansion of the Implanted Transcatheter Aortic Valve
Acronym: OptEx-TAVI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ole De Backer (Other)
Responsible Party: Sponsor-Investigator, Ole De Backer, Professor of Cardiologi, Principal investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OptEx-TAVI Trial; H-25039123 (Other: Scientific Ethics Committees for the Capital Region of Denmark)
Record Dates: First submitted 2025-06-08; First posted 2025-06-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Aortic Stenosis Disease; Valvular Heart Disease
Keywords: Aortic stenosis; Cardiovascular; Transcatheter aortic valve; Transcatheter aortic valve implantation; Valvular heart disease; TAVI
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SoC-TAVI (Active Comparator): Pre-dilatation and post-dialation optional, as per operator preference. The balloon size used for pre- or post-dilatation is left at the operator's discretion. Operators are only encouraged to post-dilate the implanted transcatheter aortic valve (TAV) in case of ≥ moderate paravalvular regurgitation or a suboptimal transvalvular gradient.
  Interventions: Procedure: SoC-TAVI
- OptEx-TAVI (Experimental): Systematic pre-dilatation and post-dilatation with an optimally-sized balloon
  Interventions: Procedure: OptEx-TAVI

INTERVENTIONS:
Procedure: OptEx-TAVI — During TAVI with either self-expanding or balloon-expandable TAVs:
  * Pre-dilatation: systematic pre-dilatation with an optimally-sized balloon.
  * Post-dilatation: systematic TAV post-dilatation with an optimally-sized balloon.
  Optimally-sized balloon:
  1. The recommended balloon size used for pre- and post-dilatation is the perimeter-derived mean diameter of the native aortic annulus minus 1 mm and should never exceed the perimeter-derived mean diameter of the native aortic annulus. A smaller-sized balloon should be considered in case of severe left ventricular outflow tract calcium and/or severely calcified leaflets in combination with a shallow sinus of Valsalva.
  2. In case of post-dilatation of the Evolut TAV (Medtronic, USA), the instructions for use (IFU) for post-dilatation of the Evolut valve should be respected.
  3. Also, a balloon-expandable TAV has to be post-dilated with an optimally-sized balloon in case of randomization to the OptEx-TAVI arm.
  Arms: OptEx-TAVI
Procedure: SoC-TAVI — During TAVI with either self-expanding or balloon-expandable TAVs: Pre-dilatation: optional, as per operator preference and post-dilatation: optional, as per operator preference. Operators are only encouraged to post-dilate the implanted TAV in case of ≥ moderate paravalvular regurgitation or a suboptimal transvalvular gradient. The balloon size used for pre- or post-dilatation is left at the operator's discretion.
  Arms: SoC-TAVI

SUMMARY:
Optimized Expansion of the implanted transcatheter aortic valve to reduce hypoattenuating leaflet thickening in non-atrial fibrillation patients undergoing transcatheter aortic valve implantation (TAVI): an international, multicentre, randomized controlled trial.

The objective is to evaluate whether TAVI with systematic optimized pre- and post-dilatation (optimized expansion (OptEx) TAVI strategy), compared to a standard of care (SoC) TAVI strategy, is superior in reducing hypoattenuating leaflet thickening as evaluated by cardiac computed tomography (CT) imaging at three months after TAVI.

The primary outcome is at least one thickened TAV leaflet involving ≥ 25% of the leaflet curvilinear dimension as assessed at cardiac CT at three months after TAVI.

DETAILED DESCRIPTION:
A total of 620 patients will be included in the OptEx-TAVI trial and randomised 1:1 to either :

* SoC-TAVI (N = 310) or
* OptEx-TAVI (N = 310)

All patients with indication for TAVI and eligible in relation to the study in- and exclusion criteria will be offered participation in the OptEx-TAVI trial.

Inclusion criteria:

* Severe symptomatic aortic stenosis patients with an indication for TAVI
* Ability to understand and to comply with the study protocol

Exclusion criteria:

* Existing indication for oral anticoagulation (e.g., atrial fibrillation, venous thromboembolism, antiphospholipid syndrome, mechanical mitral valve)
* Creatinine clearance <15 mL/min (CKD-EPI formula) or on renal replacement therapy
* Iodine contrast allergy or other condition that prohibits cardiac CT imaging

Baseline characteristics, medical history, procedural details, electrocardiogram, echocardiography and cardiac CT-scan parameters will be recorded by assessing medical charts and patient interview.

During the TAVI-procedure, patients will be treated according to randomisation to either SoC or OptEx

Planned post-procedural visits at:

* Discharge: on-site - including transthoracic echocardiography (TTE)
* 3 months visit (± 2 months): on-site - including TTE and cardiac CT scan
* 1 year (± 3 months): on-site - including TTE and cardiac CT scan
* 5 years (± 6 months): on-site - including TTE and cardiac positron emission tomography (PET)-CT scan

ELIGIBILITY:
Inclusion Criteria:

* Severe symptomatic aortic stenosis patients with an indication for TAVI
* Ability to understand and to comply with the study protocol

Exclusion Criteria:

* Existing indication for oral anticoagulation (e.g., atrial fibrillation, venous thromboembolism, antiphospholipid syndrome, mechanical mitral valve)
* Creatinine clearance <15 mL/min (CKD-EPI formula) or on renal replacement therapy
* Iodine contrast allergy or other condition that prohibits cardiac CT imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2025-10-05 (Actual); Primary Completion 2032-07-01 (Estimated); Study Completion 2033-07-01 (Estimated)

PRIMARY OUTCOMES:
At least one TAV leaflet with HALT | At three months after TAVI
  At least one TAV leaflet with hypoattenuated leaflet thickening (HALT) involving more than the base (≥ 25% of the leaflet curvilinear dimension) as assessed at cardiac CT-scan .

SECONDARY OUTCOMES:
HALT 50% | At 3 months/At 1 year
  At least one TAV leaflet with HALT involving ≥ 50% of the leaflet curvilinear dimension assessed by cardiac CT-scan
HALT 25% | At 3 months/At 1 year
  The rate of TAV leaflets with HALT involving ≥ 25% of the leaflet curvilinear dimension assessed by cardiac CT-scan
HALT 50%, multiple | At 3 months/At 1 year
  The rate of TAV leaflets with HALT involving ≥ 50% of the leaflet curvilinear dimension assessed by cardiac CT-scan
Bioprosthetic leaflet micro-calcification target-to-background ratio | At 5 years
  Ratio of bioprosthetic micro-calcification activity assessed by PET CT- scan by 18F-NaF uptake originating from the valve leaflets observed on 3 orthogonal planes after co-registration of background PET activity with contrast CT angiography.
  Only for those patients alive at 5 years and volunteering to undergo a F-NaF PET-CT-scan
Valve performance | At 3 months/At 1 year
  Intended performance of the valve (mean gradient < 20 mmHg, peak velocity < 3 m/s, Doppler velocity index ≥ 0.25, and less than moderate aortic regurgitation) by TTE as per VARC- 3 criteria
structural valve deterioration | At 5 years
  Moderate or greater hemodynamic structural valve deterioration by TTE as per VARC-3 criteria. Only for those patients alive at 5 years and volunteering to undergo a F-NaF PET-CT-scan
Bioprosthetic valve dysfunction (BVD) | At 5 years
  Severe bioprosthetic valve dysfunction (BVD) by TTE as per VARC-3 criteria. Only for those patients alive at 5 years and volunteering to undergo a F-NaF PET-CT-scan
Bioprosthetic valve failure (BVF) | At 5 years
  As per VARC-3 criteria; Only for those patients alive at 5 years and volunteering to undergo a F-NaF PET-CT-scan
Technical success | Periprocedural
  As per VARC-3 criteria
Device success | At 3 months
  as per VARC-3 criteria
Early safety | At 3 months
  As per VARC-3 criteria
Clinical efficacy | At 1 year
  As per VARC-3 criteria
Valve-related long-term clinical efficacy | At 5 years
  As per VARC-3 criteria; Only for those patients alive at 5 years and volunteering to undergo a F-NaF PET-CT-scan
Freedom from mortality | Periprocedural, at 3 months and at 1 year
  Freedom from mortality
Risk of cardiovascular mortality | At 1 year
  Risk of cardiovascular mortality. VARC-3 criteria
Risk of non-cardiovascular mortality | At 1 year
  Risk of non-cardiovascular mortality. VARC-3 criteria
Risk of acute kidney injury | At 3 months
  Risk of acute kidney injury stage 3 or 4. VARC-3 criteria
Risk of bleeding | At 3 months, 1 year and 5 years (Only for those patients alive at 5 years and volunteering to undergo a F-NaF PET-CT-scan)
  Risk of VARC-3 type 2-4 bleeding
Risk of stroke | At 3 months and 1 year
  Risk of all stroke
Risk of thomboembolism | At 5 years
  Freedom from stroke or peripheral embolism (presumably valve-related, after ruling out other non-valve aetiologies). VARC-3 criteria.
Rate of successful access | Periprocedural
  Successful access, delivery of the device, and retrieval of the delivery system
Freedom from surgery or intervention | Periprocedural and at 3 months
  Rate of freedom from surgery or intervention related to the device or to a major vascular or access-related, or cardiac structural complication
Risk of vascular complications | At 3 months
  Risk of major vascular, access-related, or cardiac structural complication, VARC-3 criteria.
Risk of aortic prosthetic regurgitation | At 3 months
  Freedom from moderate or severe aortic regurgitation. VARC-3 criteria
Risk of permanent pacemaker | At 3 months
  Risk of new permanent pacemaker due to procedure-related conduction abnormalities
Risk of procedure or valve-related hospitalization | At 1 year
  Risk of hospitalization for procedure- or valve-related causes. VARC-3

CONTACTS AND LOCATIONS:
Overall Officials: Ole De Backer, MD, PhD, FESC, Principal Investigator — The Heart Center, Rigshospitalet
Locations (10):
- Belgium (2):
  - CHU Charleroi, Charleroi
  - UZ Leuven, Leuven
- Denmark (4):
  - Skejby Hospital, Aa
  - Aalborg University Hospital, Aalborg
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense C
- Turku University Hospital, Turku, Finland
- St. Antonius Hospital, Nieuwegein, Netherlands
- Oslo universitetssygehus, Oslo, Norway
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No